CLINICAL TRIAL: NCT05103657
Title: A Phase II, 8-week-treatment, Multicenter, Randomized, Doubleblind, Placebo-controlled, Parallel Group Trial to Evaluate the Efficacy, Tolerability and Safety of Orally Administered BI 1358894 in Patients With Post-Traumatic Stress Disorder (PTSD)
Brief Title: A Study to Test Whether Taking BI 1358894 for 8 Weeks Helps Adults With Post-traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1402-0030; 2021-003154-23 (EudraCT Number)
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Post-Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — TRPC inhibitor BI 1358894

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 1358894 125 mg (Experimental)
  Interventions: Drug: BI 1358894
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1358894 — BI 1358894
  Arms: BI 1358894 125 mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is open to people aged 18 to 65 who have post-traumatic stress disorder. The purpose of this study is to find out whether a medicine called BI 1358894 improves symptoms in people with post-traumatic stress disorder.

Participants are put into 2 groups randomly, which means by chance. Participants take BI 1358894 or placebo as tablets every day for 2 months. Placebo tablets look like BI 1358894 tablets but do not contain any medicine.

Participants are in the study for about 3 months. During this time, they visit the study site about 8 times and get about 4 phone calls from the trial staff. During the study, participants answer questions in interviews and complete questionnaires so the doctors can check whether their symptoms change.

The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of Post-Traumatic Stress Disorder (PTSD) corresponding to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria
* Time since index event according to Life Events Checklist / Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Criterion A at least 3 months before screening visit
* PTSD must be the clinically pre-dominant disorder, as per investigator´s judgement. Other comorbid psychiatric disorders are allowed, unless specifically excluded in the exclusion criteria
* A total severity score of ≥ 33 on the PTSD Checklist for DSM-5 (PCL-5) at the screening visit
* Moderate to severe PTSD confirmed by CAPS-5 range ≥ 30 confirmed at screening visit
* Male or female patients, 18 to 65 years of age, both inclusively at the time of informed consent
* Women who are of child-bearing potential (WOCBP) must be able and willing to use two methods of contraception, as confirmed by the investigator, which include one highly effective method of birth control per International Council on Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1%, plus one additional barrier method
* Signed and dated written informed consent in accordance with International Council on Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Corresponding to DSM-5, had ever met diagnostic criteria for schizophrenia, schizoaffective disorder, schizophreniform disorder, bipolar disorder, delusional disorder, brief psychotic disorder or any other psychotic disorder as well as Major Depressive Disorder (MDD) with psychotic features as assessed by the Mini-International Neuropsychiatric Interview (MINI) at the time of screening
* Any psychiatric or non-psychiatric medical condition likely to negatively impact trial participation as per the judgement of the investigator
* Acute stress disorder or significant traumatic event within 3 months prior to the screening visit
* Use of stimulant medications within 3 months prior to the screening visit (Attention Deficit Hyperactivity Disorder (ADHD) diagnosis alone is not exclusionary)
* Severe traumatic brain injury (life-time) or moderate traumatic brain injury within the last 2 years prior to screening visit or 3 months for mild traumatic brain injury, based on the Ohio State University Traumatic Brain Injury (TBI) Identification Method Short Form. Or history of traumatic brain injury that would impact ability to complete trial assessments or procedures according to investigator.
* Current treatment with trauma focused therapy (i.e. Cognitive Processing Therapy (CPT), Prolonged Exposure Therapy (PE), Eye Movement Desensitization and Reprocessing (EMDR)). A psychotherapy in type, intensity and/or frequency other than trauma focused therapy is allowed if stable within the last 8 weeks prior to screening and not anticipated to change during the entire course of the trial. Long-term psychotherapy is permitted as long as patients are not in an exposure phase during the trial.
* Diagnosis of a current moderate or severe alcohol use disorder according to MINI within 3 months prior to screening visit (mild alcohol use disorder (AUD) and patients in early remission = criterion not met for between 3 & 12 months are allowed) Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- United States (37):
  - Woodland International Research Group, Inc., Little Rock, Arkansas
  - Behavioral Research Specialists, LLC, Glendale, California
  - ASCLEPES Research Centers, P.C. dba Alliance Research, Long Beach, California
  - CalNeuro Research Group Inc., Los Angeles, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, LLC, San Diego, California
  - Clinical Innovations Inc., Santa Ana, California
  - California Neuroscience Research, Sherman Oaks, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Mountain Mind. LLC, Denver, Colorado
  - CNS Clinical Research - Coral Springs, Coral Springs, Florida
  - Innovative Clinical Research, Lauderhill, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Medical Research Group of Central Florida, Orange City, Florida
  - Elixia PHC, LLC, St. Petersburg, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Emory University, Atlanta, Georgia
  - American Medical Research, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Pharmasite Research, Incorporated, Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Sisu BHR, LLC, Springfield, Massachusetts
  - NeuroBehavioral Medicine Group, Bloomfield Hills, Michigan
  - Hassman Research Institute, Berlin, New Jersey
  - Center For Emotional Fitness, Cherry Hill, New Jersey
  - Princeton Medical Institute, Princeton, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Insight Clinical Trials, Beachwood, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - The University of Texas at Austin, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Relaro Medical Trials, LLC, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Salem VA Medical Center, Salem, Virginia
- Croatia (5):
  - Clincal Hospital Centre Rijeka, Rijeka
  - Polyclinic Neuron, Zagreb
  - Solmed Polyclinic, Zagreb
  - Psychiatric Hospital 'Sveti Ivan', Zagreb
  - University Psychiatric Hospital Vrapce, Zagreb
- Finland (3):
  - Eira Medical Centre, Helsinki
  - Oulu Mentalcare Oy, Oulu
  - Mehiläinen Tampere, Tampere
- Germany (4):
  - Universitätsklinikum Aachen, AöR, Aachen
  - Zentralinstitut für seelische Gesundheit, Mannheim
  - Klinikum der Universität München - Campus Innenstadt, München
  - Universitätsklinikum Tübingen, Tübingen
- The Chaim Sheba Medical Center Tel HaShomer, Tel Litwinsky, Israel
- Mexico (4):
  - Centro para el Desarrollo de la Medicina y de Asistencia Medica Especializada S.C., Culiacán
  - Hospital Aranda de la Parra, León
  - CIT-Neuropsique S.C, Monterrey
  - BIND Investigaciones S.C., San Luis Potosí City
- Poland (3):
  - MlynowaMed, Bialystok
  - In-Vivo Sp. Z o.o., Bydgoszcz
  - MTZ Clinical Research Powered by Pratia, Warsaw
- Sweden (4):
  - Psykiatri Södra Stockholm, Enskede
  - Psykiatri Affektiva sjukdomar, Gothenburg
  - Psykiatri Sydväst Stockholm, Huddinge/Stockholm
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase II, 8-week-treatment, multicentre, randomised, double blind, placebocontrolled, parallel-group trial in patients with Post-Traumatic Stress Disorder (PTSD).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Placebo: Patients received orally, once daily for 8 consecutive weeks film-coated tablets of placebo matching BI 1358894. Placebo matching BI 1358894 was administered with water and in a consistent way, i.e. either with or without food every morning at approximately the same time.
- BI 1358894 125 mg: Patients received orally, once daily for 8 consecutive weeks 125 milligrams (mg) of BI 1358894. The dosage of 125 milligrams consisted of two film-coated tablets of 50 mg and 1 film-coated tablet of 25 mg. BI 135889 was administered with water and in a consistent way, i.e. either with or without food every morning at approximately the same time.
Period: Overall Study
Arm/Group | Placebo | BI 1358894 125 mg
Started (Randomised) | 160 | 158
Treated | 159 | 157
Completed (completed planned treatment) | 133 | 127
Not Completed | 27 | 31
Not completed — Other reasons than listed | 9 | 8
Not completed — Protocol deviation | 2 | 2
Not completed — No reason available | 5 | 4
Not completed — Burden of study procedures | 3 | 1
Not completed — Perceived lack of efficacy | 1 | 1
Not completed — Adverse Event | 6 | 14
Not completed — Not Treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): consisted of all patients that were randomised and had received at least one administration of trial drug. Patients were analysed according to the actual received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1358894 125 mg | Total
Number analyzed (Participants) | 159 | 157 | 316
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (12.9) | 42.8 (12.4) | 43.4 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 111 | 212
  Male | 58 | 46 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 35 | 64
  Not Hispanic or Latino | 130 | 122 | 252
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 10 | 16
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 26 | 72
  White | 102 | 119 | 221
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
CAPS-5 total severity score at baseline [Mean (Standard Deviation); unit: score on a scale] — Clinician-administered Post Traumatic Stress Disorder (PTSD) Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) is a 30-item clinician-administered structured interview that can be used to, make current (past month) diagnosis of PTSD and assess PTSD symptoms over the past week. The CAPS-5 as used in this trial has 20 items, each scored 0-4, to yield a score with a possible range of 0-80. Higher scores mean worse outcome.
  score on a scale | 41.3 (9.9) | 42.0 (9.6) | 41.6 (9.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered Post Traumatic Stress Disorder (PTSD) Scale for DSM-5 (CAPS-5) Total Severity Score at Week 8
Description: CAPS-5 is a 30-item clinician-administered structured interview that can be used to, make current (past month) diagnosis of PTSD and assess PTSD symptoms over the past week. Each of the 20 symptom items in the CAPS-5 is rated from 0 (absent) to 4 (extreme/incapacitating) with a single severity score combining information about frequency/amount and intensity which is yield by summing each item scores and ranges from 0 to 80 with higher scores indicating higher symptom severity. Least Squares (LS) means and confidence intervals were estimated by restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) including the fixed categorical covariates of treatment, and the stratification indicator of presence of significant childhood trauma (yes vs. no), the continuous fixed covariate of baseline CAPS-5 total severity score, time since index event (in years) and the treatment-by-visit interaction. Patient is considered as random. Unstructured covariance matrix was used.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated CAPS-5 measurements from baseline, Week 4, and Week 8. MMRM estimates of change from baseline to Week 8 is reported.
Population: Full analysis set (FAS): consisted of all patients in the treated set (TS) that had a baseline and at least one evaluable post-baseline measurement for the primary endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | BI 1358894 125 mg
Number analyzed (Participants) | 148 | 151
units on a scale | -17.19 [-19.56 to -14.81] | -17.13 [-19.52 to -14.74]
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 125 mg; Least Squares (LS) means differences and confidence intervals were estimated by REML-based MMRM including the fixed categorical covariates of treatment, and the stratification indicator of presence of significant childhood trauma (yes vs. no), the continuous fixed covariate of baseline CAPS-5 total severity score, time since index event (in years) and the treatment-by-visit interaction. Patient is considered as random. Unstructured covariance matrix was used; Test type: Other; p = 0.9726, Mixed Models for repeated measures; Mean Difference (Net) = 0.06, 95% CI 2-sided [-3.31 to 3.43] — Least Squares mean of "BI 1358894 125 mg" - Least Square mean of "Placebo"

2. Secondary Outcome: CAPS-5 Response, Defined as ≥30% CAPS-5 Reduction From Baseline at Week 8
Description: Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) is a 30-item clinician-administered structured interview that can be used to, make current (past month) diagnosis of PTSD and assess PTSD symptoms over the past week. Each of the 20 symptom items in the CAPS-5 is rated from 0 (absent) to 4 (extreme/incapacitating) with a single severity score combining information about frequency/amount and intensity which is yield by summing each item scores and ranges from 0 to 80 with higher scores indicating higher symptom severity.
  Number of participants with ≥30% CAPS-5 reduction from baseline at Week 8 is reported.
Time Frame: At baseline and at 8 weeks after start of treatment.
Population: Full analysis set (FAS): consisted of all patients in the treated set (TS) that had a baseline and at least one evaluable post-baseline measurement for the primary endpoint. Only participants with data from baseline and from Week 8 were included in the analysis of this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BI 1358894 125 mg
Number analyzed (Participants) | 129 | 129
Participants | 77 | 77
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 125 mg; Logistic regression was adjusted for fixed factors of treatment and presence of significant childhood trauma (yes vs. no); Test type: Other; p = 0.9945, Regression, Logistic; Odds Ratio (OR) = 1.002, 95% CI 2-sided [0.608 to 1.650] — BI 1358894 125 mg vs. Placebo

3. Secondary Outcome: CAPS-5 Response, Defined as ≥50% CAPS-5 Reduction From Baseline at Week 8
Description: Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5) is a 30-item clinician-administered structured interview that can be used to, make current (past month) diagnosis of PTSD and assess PTSD symptoms over the past week. Each of the 20 symptom items in the CAPS-5 is rated from 0 (absent) to 4 (extreme/incapacitating) with a single severity score combining information about frequency/amount and intensity which is yield by summing each item scores and ranges from 0 to 80 with higher scores indicating higher symptom severity.
  Number of participants with ≥50% CAPS-5 reduction from baseline at Week 8 is reported.
Time Frame: At baseline and at 8 weeks after start of treatment.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BI 1358894 125 mg
Number analyzed (Participants) | 129 | 129
Participants | 53 | 50
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 125 mg; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.7167, Regression, Logistic; Odds Ratio (OR) = 0.912, 95% CI 2-sided [0.552 to 1.504] — BI 1358894 125 mg vs. Placebo

4. Secondary Outcome: Change From Baseline on the PTSD Checklist for DSM-5 (PCL-5) Total Score at Week 8
Description: The PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (PCL-5) is a 20-item patient-reported assessment designed to measure the presence and severity of PTSD symptoms in the past month. Items on the PCL-5 correspond with DSM-5 criteria for PTSD. Each item is rated on a five point Likert scale, from 0 (not at all) to 4 (extremely) yielding a total score from 0-80 with higher scores indicating higher severity of the symptoms.
  Least Square (LS) means and confidence intervals were estimated by restricted maximum likelihood (REML)-based mixed model repeated measures (MMRM) including the fixed categorical covariates of treatment, and the stratification indicator of presence of significant childhood trauma (yes vs. no), the continuous fixed covariate of baseline CAPS-5 total severity score, time since index event (in years) and the treatment-by-visit interaction. Patient is considered as random. Unstructured covariance matrix was used.
Time Frame: The MMRM model is a longitudinal analysis and it incorporated PCL-5 measurements from baseline, Week 4, and Week 8. MMRM estimates of change from baseline to Week 8 is reported.
Population: Full analysis set (FAS): consisted of all patients in the TS that had a baseline and at least one evaluable post-baseline measurement for the primary endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | BI 1358894 125 mg
Number analyzed (Participants) | 148 | 151
units on a scale | -19.21 [-21.80 to -16.61] | -18.55 [-21.12 to -15.98]
Statistical Analysis 1: Comparison: Placebo vs BI 1358894 125 mg; Least Square (LS) means differences and confidence intervals were estimated by REML-based MMRM including the fixed categorical covariates of treatment, and the stratification indicator of presence of significant childhood trauma (yes vs. no), the continuous fixed covariate of baseline CAPS-5 total severity score, time since index event (in years) and the treatment-by-visit interaction. Patient is considered as random. Unstructured covariance matrix was used; Test type: Other; p = 0.7230, Mixed Models for Repeated Measures; Mean Difference (Net) = 0.66, 95% CI 2-sided [-3.00 to 4.32] — Least Square mean of "BI 1358894 125 mg" - Least Square mean of "Placebo"

ADVERSE EVENTS:
Time Frame: "All-Cause Mortality" "Serious Adverse Events" and "Other Adverse Events": From first administration of BI 1358894 or placebo to last administration of BI 1358894 or placebo + 4 weeks of residual effect period, up to 13 weeks.
Description: Treated Set (TS): consisted of all patients that were randomised and had received at least one administration of trial drug. Patients were analysed according to the actual received treatment.
Arm/Group | Placebo | BI 1358894 125 mg
All-Cause Mortality (participants affected / at risk) | 1/159 | 0/157
Serious Adverse Events (participants affected / at risk) | 10/159 | 12/157
Other Adverse Events (participants affected / at risk) | 38/159 | 56/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | BI 1358894 125 mg (N=157)
Haematochezia (Gastrointestinal disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amnesia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 1
Suicidal ideation (Psychiatric disorders) | 4 | 4
Suicide attempt (Psychiatric disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | BI 1358894 125 mg (N=157)
Nausea (Gastrointestinal disorders) | 15 | 7
Fatigue (General disorders) | 2 | 10
Weight increased (Investigations) | 3 | 11
Increased appetite (Metabolism and nutrition disorders) | 2 | 8
Dizziness (Nervous system disorders) | 8 | 12
Headache (Nervous system disorders) | 20 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/57/NCT05103657/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT05103657/SAP_001.pdf